CLINICAL TRIAL: NCT03007017
Title: Novel Strategies for Innovating Deceased Donor Procurement
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Maryland, Baltimore (Other)
Collaborators: Living Legacy Foundation (Unknown)
Responsible Party: Principal Investigator, Joseph Scalea, Assistant Professor of Surgery Director of Pancreas and Islet Cell Transplantation, University of Maryland, Baltimore
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 00071879
Record Dates: First submitted 2016-12-08; First posted 2016-12-30 (Estimated); Last update posted 2021-06-09 (Actual); Status verified 2021-06

CONDITIONS: Kidney Failure, Chronic
MeSH Terms: conditions — Kidney Failure, Chronic | interventions — Standard of Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Arm 1 (Experimental): Patients selected for this arm will receive the left kidney from the new method of organ retrieval.
  Interventions: Procedure: Deceased donor nephrectomy, prior to cross clamp of donor aorta
- Arm 2 (Active Comparator): Patients selected for this arm will receive the normal standard of care operational kidney from retrieval.
  Interventions: Procedure: Deceased donor nephrectomy, standard of care

INTERVENTIONS:
Procedure: Deceased donor nephrectomy, prior to cross clamp of donor aorta — The investigators will perform a prospective investigation of organ recoveries during which the left kidney will be removed prior to cessation of cardiac activity. The second kidney will be removed in the standard fashion. To do this, investigators will adopt techniques used in living donor kidney transplantation. Specifically, a specialized vascular stapler will be used to divide the renal artery at the level of aorta, followed by the vein, at the level of the vena cava. As such, no "cuff" of abdominal aorta or vena cava will be present on the target kidneys. Once removed from the body, just as is done for living donor kidney transplantation, the kidneys will be immediately flushed. As this ex-vivo flush is already performed for cadaveric kidney transplantation, there should be no additional cost for performing this portion of the procedure. Approximately 15 minutes of additional surgical dissection (prior to stopping the heart) will be required under the proposed study.
  Arms: Arm 1
Procedure: Deceased donor nephrectomy, standard of care — The investigators will remove the right kidney in the stand of care procedures for cadaveric kidney transplantation
  Arms: Arm 2

SUMMARY:
Despite many efforts to increase the size of the donor pool, there is a large and growing disparity between the number of donor kidneys available for transplantation and the number of patients on the transplant waiting list. Increasing the quality of currently available donor kidneys would potentially improve the longevity of deceased donor kidney transplants by years, thus increasing the rate of transplantation patients on the kidney transplant waiting list. In addition, recipients of higher quality kidneys have shorter hospital stays and lower total hospital charges. By innovating the organ donation process, such that deceased donor kidneys are removed prior to the cessation of cardiac activity, rather than after, it may be possible to improve the quality of the kidney before transplantation, resulting in improved function after transplantation and increased longevity of these transplanted kidneys. Further, this improved kidney quality is highly likely to translate to reduced need for renal dialysis and other high-cost interventions, yielding lower total hospital charges. In this study we will test the hypothesis that, through a cost-free technical innovation, the quality of deceased donor kidneys could be improved significantly, saving thousands more lives per year and reducing total health care expenditures on renal transplantation.

ELIGIBILITY:
Inclusion Criteria:

1. Currently listed to receive a deceased donor kidney transplant
2. Able to fully understand the informed consent document
3. Recipient over the age of 18 years

Exclusion Criteria:

1. Recipients undergoing a bilateral native nephrectomy at time of transplant
2. Recipients undergoing dual (liver-kidney, kidney-pancreas, pediatric en bloc) transplant
3. Individuals who are unable to understand the informed consent document
4. Recipient under age 18 years
5. Recipients receiving desensitization protocols for high levels of donor specific antibodies

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2017-01 (Actual); Primary Completion 2021-06-07 (Actual); Study Completion 2021-06-07 (Actual)

PRIMARY OUTCOMES:
Sequence of organ procurement | 1 year
  Renal allograft survival
Kidney quality | 3 months
  Incidence of delayed renal graft function

CONTACTS AND LOCATIONS:
Locations (1):
- University of Maryland, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No